CLINICAL TRIAL: NCT04076098
Title: Efficacy of Locally Delivered Minocycline in Advanced Periodontitis. A Clinico-microbiological Study
Brief Title: Locally Delivered Minocycline in Advanced Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahsa University (Other)
Responsible Party: Principal Investigator, Professor. Dr. Tara Bai Taiyeb Ali, Professor, Mahsa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP139-02/18
Record Dates: First submitted 2019-08-02; First posted 2019-09-03 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Periodontitis, Adult
MeSH Terms: conditions — Chronic Periodontitis | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minocycline (Experimental): Minocycline gel
  Interventions: Drug: Minocycline Hydrochloride
- Placebo (Placebo Comparator): Similar gel without the active agent
  Interventions: Drug: Minocycline Hydrochloride

INTERVENTIONS:
Drug: Minocycline Hydrochloride — Administration of Periocline gel into the periodontal pockets will be carried out until it overflows the pockets
  Other Names: Periocline

SUMMARY:
Local drug delivery provides higher concentrations in the availability of the drug at the specific infected sites with the advantage of sustained release. Periocline is a long acting , sustained release local drug delivery system consisting of 2% minocycline hydrochloride in an ointment containing microcapsule type particles. Periocline contains 20mg of minocycline in 0.5 gm of gel in a disposable polypropylene applicator (2% minocycline HCl).

Research has yielded promising results with the local application of minocycline in the treatment of periodontal disease, compared with other non-surgical therapies. However, there is scarcity of reports on the use of local delivery agents with respect to new range of putative pathogens in advanced periodontitis, wherein the tissue invasive anaerobic organisms are present and possibly compromised host response, hence resulting in an exaggerated breakdown of periodontal tissues at the affected sites. The effect of Minocycline on new putative pathogens, such as Filifactor alocis and oral phylotypes of phyla Synergistetes and TM7 (referred to hereafter as oral Synergistetes and oral TM7s), has not been investigated yet.

Hence, the aim of the present study is to evaluate the efficacy of a local delivery agent containing minocycline (Periocline, Sunstar, Japan) as an adjunct to SRP in the treatment of deep periodontal pockets around teeth in advanced periodontitis and the antimicrobial effect on the red complex and the new putative pathogens.

DETAILED DESCRIPTION:
The subjects for this randomized controlled, parallel arm study will be selected from the primary health care in the Faculty of Dentistry, MAHSA University. In this clinical trial, 50 patients with advanced periodontitis will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* systematically healthy patients with age range between 20- 60 years,
* diagnosed with untreated Advanced Periodontitis with a pocket depth ≥6mm around two or more teeth, in two or more quadrants.

Exclusion Criteria:

* Patients given antibiotics or anti-inflammatory drugs in the past 6 months,
* allergic to tetracycline,
* pregnant or nursing females,
* those using chlorhexidine or any other mouth rinse

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Change in Probing pocket depth (PPD) | baseline to 12 weeks
  Periodontal pocket is measured from the gingival margin to the base of the periodontal pocket using a UNC periodontal probe (which is graduated from 1mm to 15mm). The measurement of periodontal pocket depth is a continuous scale. PPD is taken at 6 points on each tooth. The mean of the PPD will be obtained for each patient and subjected to statistical analysis.
Change in the numbers of Periodontal pathogens | baseline to 12 weeks
  Plaque samples taken from periodontal pockets on paper points will be first stored and later analysed for the presence and number of periopathogens using quantative Polymerase Chain Reaction (q-PCR).
  The following periodontal pathogens will be assessed:
  * Red complex (Porphyromonas gingivalis, Tannerella forsythia,and Treponema denticola)
  * Filifactor alocis,
  * oral phylotypes of phyla Synergistetes
  * Phylum TM7
Clinical Attachment Levels (CAL) | baseline, 6 weeks and 12 weeks
  change in CAL

SECONDARY OUTCOMES:
Plaque Index | baseline to 12 weeks
  change in Plaque scores (Silness and Loe Plaque index, 1964) The score ranges from 0-3 and it is a continuous scale. '0' - no plaque '1' - thin plaque which is not visible by naked eye '2' - Moderate accumulation plaque seen by naked eye '3' - abundance of plaque.
  Calculation total score /number of surfaces examined = Index score for each patient. Mean plaque score is calculated for all the patients.
Bleeding Index | baseline to 12 weeks
  change in Bleeding scores (Papillary bleeding index, Muehlemann 1977) The score ranges from 0-4 and it is a continuous scale. '0' - no bleeding '1' - Single discrete bleeding point '2' - Single line of blood appears '3' - Interdental papilla fills with blood after probing '4' - profuse bleeding after probing
  Calculation total score /number of surfaces examined = Index score for each patient. Mean plaque score is calculated for all the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Taiyeb Ali, MSc, FDSRCS, Principal Investigator — Mahsa University
Locations (1):
- MAHSA University, Jenjarum, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No